

# **Trial Protocol**

A randomised controlled trial of the prediction of diminutive/small polyp histology: a comparison between didactic training versus self-directed computer based training

This protocol has regard for the HRA guidance

# Protocol development and sign off

As per EC guidance (ENTR/CT2) the protocol should be signed by the CI and by the Sponsor to confirm approval of the protocol. NOTE: For UoB sponsored trials, the sponsor will confirm approval of the protocol by signing the IRAS form and therefore a signature on the protocol is not required. The sponsor must be notified of all amendments to the protocol, both substantial and nonsubstantial. Review of amendments by the sponsor will act as the confirmation that the sponsor confirms approval of the amended protocol.

# **Key Protocol Contributors**

| The following people have contributed to the writing of this protocol: | |
|---|---|
| Name: | Affiliation and role: |
| Dr Samuel Smith | Clinical research fellow, Institute of Translational Medicine |
| Dr Marietta lacucci | Reader in gastroenterology, Institute of Translational Medicine |
| Hollie Caulfield | Research co-ordinator, Institute of Translational Medicine |

# **Protocol Amendments**

| The following amendments and/or administrative changes have been made to this protocol since the implementation of the first approved version | | | | |
|---|---|---|---|---|
| Amendment<br>number | Date of amendment | Protocol<br>version<br>number | Type of amendment | Summary of amendment |

2 of 27 Training Module Version number: 1.0 Version date: 09/01/2018 Page:

# CI Signature Page

The undersigned confirm that the following protocol has been agreed and accepted and that the Chief Investigator agrees to conduct the trial in compliance with the approved protocol and will adhere to the principles outlined in the Medicines for Human Use (Clinical Trials) Regulations 2004 (SI 2004/1031), amended regulations (SI 2006/1928) and any subsequent amendments of the clinical trial regulations, GCP guidelines, the Sponsor's SOPs, and other regulatory requirements as amended.

I agree to ensure that the confidential information contained in this document will not be used for any other purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of the Sponsor.

I also confirm that I will make the findings of the study publically available through publication or other dissemination tools without any unnecessary delay and that an honest accurate and transparent account of the study will be given; and that any discrepancies from the study as planned in this protocol will be explained This protocol has been approved by:

**Trial Name:** Diminutive training module: didactic training versus computer based self-

learning- a multicentre international study

**Protocol Version Number:** Version: 1.0

**Protocol Version Date:** 09/01/2018

CI Name: Dr Marietta Iacucci

Trial Role: **Chief Investigator** 

Signature and date:

# Sponsor statement:

Where the University of Birmingham takes on the sponsor role for protocol development oversight, the signing of the IRAS form by the sponsor will serve as confirmation of approval of this protocol.

Training Module Version number: 1.0 Version date: 09/01/2018 Page:

Training Module Version number: 1.0 Version date: 09/01/2018 

# Administrative Information

Use this page to document the key contact personnel for the trial.

| Sponsor | |
|---|---|
| University of Birmingham | 0121 414 7618 |
| Sponsor contact: Dr Sean Jennings | researchgovernance@contacts.bham.ac.uk |
| Research Governance Team | |
| University of Birmingham | |
| Birmingham, B15 2TT | |

| Chief Investigator | |
|-------------------------------------|----------------------------|
| Dr Marietta Iacucci | Reader in gastroenterology |
| Institute of Translational Medicine | 0121 3718026 |
| University of Birmingham | m.iacucci@bham.ac.uk |
| Birmingham, B15 2TT | |

| Sponsor's Medical Expert for the Trial | |
|----------------------------------------|----------------------------|
| Dr Marietta Iacucci | Reader in gastroenterology |

| Research fellow | |
|---|---|
| Dr Samuel Smith | Clinical research fellow |
| Institute of Translational Medicine University of Birmingham Birmingham, B15 2TT | 0121 3718026<br>s.c.l.smith@bham.ac.uk |
| Co-investigator | |
| Dr John Saltzman | Gastroenterologist |
| Brigham and Women's Hospital<br>Boston, USA | JSALTZMAN@PARTNERS.ORG |
| Co-investigator | |
| Jennifer Nayor | |
| Brigham and Women's Hospital<br>Boston, USA | jnayor@bwh.harvard.edu |
| Co-investigator | |
| Dr David Greenwald | Gastroenterologist |
| New York, USA | david.greenwald@mountsinai.org |

Training Module Version number:1.0 Version date: 09/01/2018 

| Co-investigator Co-investigator | |
|---------------------------------|---------------------------------|
| Dr Toshio Uraoka | Gastroenterologist |
| Tokyo, Japan | toshi_urao@yahoo.co.jp |
| Co-investigator | |
| Dr Takayaki Matsumoto | Gastroenterologist |
| Tokyo, Japan | t.matsu.1215@i.softbank.jp |
| Co-investigator | |
| Co-investigator | |
| Dr Cristina Trovato | Gastroenterologist |
| Milan, Italy | cristina.trovato@ieo.it |
| Co-investigator | |
| Dr Valentina D'Angelo | Gastroenterologist |
| Napoli, Italy | |
| | <u>'</u> |
| Co-investigator | |
| Dr Timo Rath | Gastroenterologist |
| Germany | <u>Timo.Rath@uk-erlangen.de</u> |
| Co-investigator | I |

| Trial Office Contact Details | |
|-------------------------------------|--------------------------|
| Hollie Caulfield | Research co-ordinator |
| Institute of Translational Medicine | 0121 3718182 |
| University of Birmingham | h.k.caulfield@bham.ac.uk |
| Birmingham, B15 2TT | |


# **Trial Summary**

#### **Title**

A randomised controlled trial of the prediction of diminutive/small polyp histology: a comparison between didactic training versus self-directed computer based training

### **Background**

Colonoscopy is the gold standard for detection of colonic polyps and colorectal cancer. Novel endoscopic enhancement by virtual electronic chromoendoscopy such as narrowband imaging [NBI, Olympus, Japan], Fuji Intelligent Chromo Endoscopy [FICE, Fujifilm, Japan], i-scan [Pentax, Japan], techniques have been developed to aid endoscopists to better characterize colonic polyps and predict histology thus facilitating the adoption of the new paradigm of resect and discard i.e. the PIVI-ASGE strategy resulting in cost savings and avoidance of complications in patients. Several training modules have been developed and used in prior studies evaluating the performance of endoscopic image-enhancement technologies. Different training methods, have been evaluated and include face-to-face, interactive didactic teaching or web-based/computer-based self-learning teaching modules. The superiority of one training method over the other has not been well evaluated.

# **Trial Design**

Multi-centre, international randomised controlled trial

# Methodology

# **Participant Population**

Participants will be consultants (gastroenterologists or surgeons) who are experienced in colonoscopy, training gastroenterologists, nurse endoscopists and junior doctors/medical students (who are naive in colonoscopy).

We aim to recruit 10-20 consultants/attending, 10-20 trainees/GI fellows, 10-20 nurse endoscopists (if applicable) and 10-20 junior doctors (non-GI trainees) from each centre. The participants will be randomised to receive self-directed computer based learning or face-to-face classroom didactic computer training module.


The above will be replicated at other centres: UK, USA, Italy, Germany and Japan.

Study duration: 2 years

# **Statistical Methodology**

Performance characteristics of the participants for diagnosing colonic neoplastic vs. non neoplastic lesions (sensitivity, specificity, NPV, PPV and accuracy) will calculated by comparing predicted histology with actual histology for all polyps and for those diagnosed with high confidence.. These performance characteristics between the two groups (face-toface classroom training vs. self training module) will be compared using the Fisher's ex- act test. A P value of <0.05 will be considered to be statistically significant. Kappa statistic will be used to determine inter-observer agreement in polyp video classification during the training session.

# Sample size

Assuming a non-inferiority trial with one-sided distribution (face to face training versus computer based training), and power of 90% the sample size is 375 observations (observation=1 video scored). This falls to 271 observations if 0.80 1-beta error is set. As we will use 60 videos per participants, we would need a minimum of 7 participants in each centre. To minimise any potential errors we aim to recruit 10-20 participants from each group (as described above) from each centre.

# **Objectives**

To assess the impact of didactic face-to-face training vs. self-directed computer based training module.

To evaluate the impact of an educational training module has on the ability of clinicians to differentiate small/diminutive polyps.

### **Outcome Measures**

A pre-training assessment will be completed by participants. Performance at predicting histology (neoplastic vs. non-neoplastic) will be assessed using sensitivity, specificity, PPV, NPV and accuracy. The proportion of high and low confidence diagnoses will be also documented.

8 of 27 Version date: 09/01/2018 Page:

Following training, participants will immediately complete a post-training assessment and performances will be observed comparing with pre-training assessment. A follow up assessment at 6 months will be completed to assess the retention and sustainability of skills acquired.

Kappa inter-observer variability between the raters will be assessed.

# Intervention

Training module: didactic face-to-face classroom training or computer-based selflearning training module

9 of 27 Training Module Version number:1.0 Version date: 09/01/2018 Page:

### **Trial Schema**

Participants will be invited to attend educational eventidentified from local hospitals and regional training groups

Participants agree to take part

Novice endoscopists (junior doctors/medical students below registrar level, gastroenterology trainees (GI fellows), nurse endoscopists

Consultants/attending (experienced colonoscopists)

Participants complete pre-training assessment-72 videos (24 NBI, 24 iScan, 24 BLI, 2 weeks before training)

Participants randomised to either didactic training or computer based selflearning

Didactic training from an expert endoscopists

Computer-based self-learning

Post-training assessment 72 videos (24 NBI, 24 iScan, 24 BLI,)) within 72 hours of training

3-4 months: Participants to complete a further assessment


# **Table of Contents**

| Prot | tocol development and sign off | 2 |
|---|---|---|
| Key | Protocol Contributors | 2 |
| Dr S | Samuel Smith | 2 |
| Dr N | Marietta lacucci | 2 |
| Holl | llie Caulfield | 2 |
| Prot | tocol Amendments | 2 |
| CI Si | Signature Page | 3 |
| Spor | onsor statement: | 3 |
| Adm | ministrative Information | 5 |
| Trial | al Summar | 7 |
| Title | le | 7 |
| | ninutive polyp training module using novel endoscopic imagin: a comparison between d self-directed computer based training | |
| Tria | al Design | 7 |
| Obje | jectives | 7 |
| Part | rticipant Population and Sample Size Error! Boo | okmark not defined. |
| Out | tcome Measures | 8 |
| Inte | ervention Error! Boo | okmark not defined. |
| Tria | al Schema | 10 |
| Tabl | ole of Contents | 11 |
| 1. | Background and Rationale | 13 |
| 1.1. | . Trial Rationale | 16 |
| 1.2. | Justification for participant population | 16 |
| 1.3. | Justification for design | 17 |
| 2. | Aims, Objectives and Outcome Measures | 17 |
| 2.1. | . Aims and Objectives | 17 |
| 2.2. | Outcome Measures | 17 |
| 3. | Trial Design and Setting | 17 |
| 3.1. | Trial Design | 17 |
| 3.2. | Trial Setting | 17 |
| 4. | Eligibility | 17 |
| 4.1. | . Inclusion Criteria | 17 |
| 4.2. | Exclusion Criteria | 18 |
| 5. | Recruitment, Consent, Enrolment and Randomisation | 18 |
| 5.1. | . Recruitment | 18 |
| 5.2. | Consent | 18 |

| 5.3. | Randomisation | 18 |
|--------|-----------------------------------------|---------------------------|
| 5.4. | Blinding | 18 |
| 6. | Trial procedures and assessments | 19 |
| 6.1. | Summary of assessments | 19 |
| 6.2. | Schedule of Assessments | 19 |
| 7. | Data Handling and Record Keeping | 19 |
| 7.1. | Source Data | 19 |
| 7.2. | CRF CompletionErro | or! Bookmark not defined. |
| 7.3. | Data Management | 20 |
| 7.4. | Archiving | 20 |
| 8. | End of Trial Definition | 20 |
| 9. | Statistical Considerations | 20 |
| 9.1. | Statistical Analysis | 20 |
| 9. | .1.1. Planned Randomisation Methodology | 21 |
| 9. | .1.2. Planned Sub Group Analyses | 21 |
| 9. | .1.3. Planned Final Analyses | 21 |
| 9. | .1.4. Power Calculations | 21 |
| 10. | Trial Organisational Structure | 21 |
| 10.1 | L. Sponsor | 21 |
| 10.2 | 2. Trials Office | 22 |
| 11. | Confidentiality and Data Protection | 22 |
| 12. | Insurance and Indemnity | 22 |
| 13. | Access to the final trial dataset | 22 |
| 14. | Publication Policy | 22 |
| 15. | Reference ListReferences: | 22 |
| A none | andiaa | 25 |

# 1. Background and Rationale

Colonoscopy is the gold standard for screening for bowel cancers and detection of precursors to colorectal cancer (polyps). Early detection of polyps, allows endoscopic removal and therefore reduction in colorectal cancer. With improvements in technology endoscopists are detecting more lesions within the bowel with the majority small/diminutive <5mm (80%). however the clinical relevance of these lesions is minimal as the risk of advanced histology or cancer is <1%1,2,3. The current practice involves removing these lesions and sending for histopathological assessment, incurring a significant risk to the patient, cost and is timeconsuming, with very little benefit<sup>4,5</sup>. Novel imaging techniques including Narrow-band imaging (NBI-Olympus, Japan), i-Scan Optical enhancement (OE-Pentax, Japan) and Bluelight laser imaging (BLI- Fujifilm, Japan) can help endoscopists characterise these small lesions between being neoplastic and non-neoplastic (hyperplastic) 6,7,8,9. NBI involves the narrowing of bandwidths of light using a light filter. The light at this end of the spectrum is absorbed by haemoglobin (protein found within blood) therefore making blood vessels more pronounced. During the process whereby a polyp develops and later becomes neoplastic, there is an increase in blood vessels compared with normal tissue or hyperplastic polyps (benign), therefore NBI can be used to detect such lesions <sup>10,11</sup>. I-Scan OE is an alternative imaging technique which enhances the pattern of the surface of polyps as well as the blood vessels, by manipulating dark-light borders and red, blue and green components of light. Blue laser imaging (BLI) is also new system for image-enhanced endoscopy using laser light. Blue laser imaging utilizes two monochromatic lasers (410 and 450 nm) instead of xenon light. A 410 nm laser visualizes vascular microarchitecture, similar to narrow band imaging, and a 450 nm laser provides white light by excitation.

These novel technologies have been demonstrated to be superior over standard white light endoscopy with NBI the most extensively investigated. A systematic analysis of 6 studies >500 polyps, resulted in a pooled sensitivity of 92%, spec 86%, accuracy of 89% at differentiating neoplastic from non-neoplastic lesions when using NBI <sup>12</sup>. Head to head studies of NBI versus white light endoscopy (WLE) have shown NBI is better at differentiating between neoplastic and non-neoplastic lesions <sup>10, 13, 14</sup>. Similar results have been found with i-Scan, with performances better than WLE and like NBI are similar to chromoendoscopy (a technique that involves spraying dye over bowel mucosa which is time-consuming and costly) <sup>15, 16</sup>. BLI is a newer imaging platform, with the current evidence suggesting it is effective at differentiating polyps (neoplastic versus non-neoplastic) with


accuracies of 95.2%<sup>17</sup>, and when comparing with white light endoscopy the miss rate of adenoma was significantly lower with BLI (1.6% versus 10.0% p=0.001)<sup>18</sup>.

In order to characterise between neoplastic and non-neoplastic lesions, endoscopic scoring systems have been developed to assist endoscopists. Examples include NICE (NBI International Colorectal Endoscopic)<sup>3</sup> (Appendix 1).

Recently lacucci et al. have developed a simplified classification system (SIMPLE- Simplified Identification Method for Polyp Labelling during the Endoscopy) for optical diagnosis of small and diminutive adenomas, SSA/Ps and hyperplastic polyps using the newly introduced OE-iSCAN system which achieved a high degree of diagnostic accuracy for small/diminutive polyp diagnosis. Furthermore, they have showed that a training module on SIMPLE classification resulted in an overall NPV of 91.3% <sup>19</sup>. This user-friendly classification system can be used by experienced and non-experienced gastroenterologists on multiple endoscopy imaging platforms to differentiate neoplastic from non-neoplastic polyps (Appendix 1). A classification system developed by Bisschops R et al recently using BLI called BASIC (BLI Adenoma Serrated International Classification). This takes into account the polyp surface, pit appearance and vessels, which has shown to have a high concordance amongst experts<sup>20</sup>.

In the hands of experts using NBI-NICE classification system accuracies of 98.9%, sensitivity 98%, specificity 100%, NPV 97.7% and PPV100% were demonstrated when diagnosis was made with high confidence. Essential to the adopted use of these classifications is training for endoscopists, both experienced and those in training. There is good evidence that there is a short learning curve involved when using NBI<sup>21</sup>. One study using a self-administered computer based training module, community based gastroenterologists (non-expert) were able to reach excellent NPV of >90% but fell short of other requirements (prediction of surveillance intervals) <sup>22</sup>. Much like NBI, the learning curve at acquiring the skills in order to differentiate between hyperplastic and adenomatous lesions using i-Scan has been investigated. An early study by Neumann et al demonstrated a rapid learning curve with 4 endoscopists without previous experience with i-scan reached an accuracy of at least 85% after reviewing 67-110 lesions (with individualised feedback) following a 1 hour teaching session on pit pattern analysis<sup>23</sup>.

There have attempts at identifying the most effective training tool and method at teaching non-experts how to characterise lesions effectively. Studies have used still images of lesions<sup>24</sup>,


however this is limited as it does not reflect real-life practice as it does not allow views from different angles. It is thought videos simulate real-life practice as close as possible. A study using videos has demonstrated trainees were able to achieve accuracies of 90%<sup>25</sup>.

More recently Rastogi's group sought to identify which training method was more effective in prediction of diminutive polyp histology amongst trainees: didactic face to face training versus computer-based self-learning <sup>26</sup>. The participants were randomised to either receive didactic training in the form of a classroom training session or self-learning via computer-based material on characterisation of polyps using NBI. Trainees reviewed 40 videos of diminutive polyps with the histology being revealed and explained. Both groups were given a further 40 videos for testing. This study found those taught in the didactic group characterised polyps with higher confidence, but the overall performance was similar in the two groups. The accuracy and sensitivity were slightly better in the self-learning group (93.9% vs 85.7% p 0.01 and 95.0% vs 86.9%; p0.03 respectively) in those polyps assessed with high confidence. This study demonstrates that a computer-based training module can be as effective in didactic training, perhaps a reflection on the amount of online self-learning trainees are exposed to.

We aim to recruit participants to receive either didactic face-to-face training or self-directed computer based learning, whereby participants will be taught how to characterise lesions using the NICE, BASIC and SIMPLE classification. We aim to recruit trainees, novice endoscopists and experienced endoscopists to compare the different groups. Pre- and post-training assessments will be completed allowing us to examine the impact of training, which will consist of 40-60 videos (equal proportion of NBI, iScan OE and BLI) in the pre-training assessment and 40-60 videos (different set of videos but also equal proportion of NBI, iScan OE and BLI) in the post-training assessment. A follow up assessment will be completed at 6 months to assess the retention of skills and sustainability of colonic polyp characterisation using the optical diagnosis techniques. An existing library of NBI and OE-iScan videos will be used and further videos will be collected during routine colonoscopies with patients consenting for images to be used for teaching purposes.


### 1.1. Trial Rationale

We hypothesise that following the training module there will be an improvement in performance between the pre-training and post-training assessments. We also hypothesise that there will be no difference between the didactic face-to-face group and the self-training group.

This is an important study as better characterisation of small polyps may eventually lead to a 'resect and discard' strategy in the future. This involves characterising small or diminutive polyps (<10mm) as either non-neoplastic or neoplastic, resecting the lesion but not sending for histopathological analysis, which has significant cost savings. In order to do this training is essential. Whilst didactic training is attractive, it is costly and resource heavy. The option of self-directed learning is an attractive one as it can be delivered at times that suit the user, at their pace and can be delivered in greater volumes.

This study is unique as it is examining the impact of the training module on different groups of participants (novice, training and experienced endoscopists), using multiple endoscopic platforms(NBI, i-Scan OE and BLI) at a multicentre, international level. It will enable us to assess whether the training module improves performance using different imaging modalities.

# 1.2. Justification for participant population

The participants included will be those that will need better polyp characterisation in everyday endoscopic practice, so they are ideal candidates. Novice endoscopists will be invited to examine the effect of the training module on participants without previous experience.

16 of 27 Training Module Version number: 1.0 Version date: Page:

### 1.3. Justification for design

The training module will be carried out on the same day as the post-training assessment, in order to avoid any bias with erosion of knowledge/skills over time.

# 2. Aims, Objectives and Outcome Measures

# 2.1. Aims and Objectives

Hypothesis: performances at predicting the histology of small/diminutive polyps improves following both the didactic face-to-face feedback training and self-directed computer based training. We also hypothesise that there will no overall difference between the two teaching groups.

### 2.2. Outcome Measures

Outcome measures will include accuracy of polyp prediction, sensitivity, specificity, positive predictive value and negative predictive value. Proportion of high confidence diagnoses will also be recorded. Kappa statistics will be used to determine interobsever agreement in polyp video classification.

# 3. Trial Design and Setting

# 3.1. Trial Design

A multi-centre international randomised controlled trial.

# 3.2. Trial Setting

University of Birmingham/academic setting, plus other international centres (UK, USA, Japan, Italy, Germany)

# 4. Eligibility

### 4.1. Inclusion Criteria

- Experienced colonoscopists: fully independent and have completed >1000 procedures
- Nurse endoscopists: fully independent colonoscopists (if applicable)
- Training colonoscopists: gastroenterology trainee in the process of training in colonoscopy
- Novice colonoscopists: junior doctors/medical students who have no experience of colonoscopy


### 4.2. Exclusion Criteria

Inability to consent to take part in the study.

# 5. Recruitment, Consent, Enrolment and Randomisation

#### 5.1. Recruitment

Participating centres will be identified by the chief investigator (MI) and co-investigator (SS). Potential participants will be approached via email via lead investigators from each centre. Once participants have agreed to take part they will be randomised using sealed envelope software/Microsoft excel). No patient records will be accessed for the purposes of this study.

#### 5.2. Consent

Consent to collect data, store the information at the University of Birmingham and publish the final data collected will be sought from all participants online prior to the collection of the preand post-training assessment.

The videos used will not contain any patient identifiable information and consent for their use for educational purposes has already been sought via a written consent form and have been used in other studies.

#### 5.3. Randomisation

Participants will be randomised into either didactic face-to-face training or computer selftraining module. This will take place prior to the training event and participants will be informed of which group they have been allocated on the day by using a computerized stratified randomisation sequence where a computer-generated random number will be assigned to each participant and then randomized to each arm to ensure a balanced number in both groups.

### 5.4. Blinding

Due to the nature of the intervention, participants cannot be blinded.

18 of 27 Version date: 09/01/2018 Page:

# 6. Trial procedures and assessments

# 6.1. Summary of assessments

| | Enrolment | Allocation |
|---------------------------|----------------------|------------|
| TIMEPOINT** | At teaching sessions | |
| Eligibility screen | Х | |
| Informed consent | Х | |
| INTERVENTIONS: | | |
| [Didactic training] | х | |
| [Computer based training] | х | |

#### 6.2. Schedule of Assessments

Participants who agree to take part in the study will complete a pre-training assessment prior to the training day. Assessment material will be uploaded on REDCap, hosted via the University of Birmingham. Each participant will receive a link via email to complete the assessments. Each participant will be asked to assess: Quality of video High/Low, NICE classification, SIMPLE classification, BASIC classification, High/Low confidence and Hazewinkel criteria for each video. This will be completed at least 2 weeks prior to the training day. On the training day participants will receive either didactic face-to-face feedback training or computer-based training (identical). A post-training assessment will be completed within 72 hours of training (same videos as pre-training but in a different randomised order). The website will self-populate the data in Microsoft Excel documents. Participants will then be invited to complete a final assessment at 3-4 months, which will conclude the study.

# 7. Data Handling and Record Keeping

# 7.1. Source Data

19 of 27 Training Module Version number:1.0 Version date: 09/01/2018 Page:

The source data will be completed directly on to the forms provided to participants. This will include:

Experience: number of colonoscopies in lifetime/year, experience with NBI/iScan OE/BLI, stage of training if applicable.

Excel spreadsheets will be utilised to enter: quality of video (low/high), NICE (adenoma, hyperplastic polyp, invasive carcinoma), SIMPLE (hyperplastic, SSA, adenoma) and Hazewinkel criteria for SSA, and high/low confidence prediction.

# 7.2. Data Management

Data will be collected on Microsoft excel via canvas.bham.ac.uk. Participants will be allocated an ID number (centre initials followed by participant initials). This will be anonymised.

### 7.3. Archiving

Data collected during this study, will be kept in locked filing cabinet at all times, any online data that is received will be stored on a secure system, which only the study team will have access too. The data will be stored for use until the findings and paper are written. After this time, it will be archived for a minimum on 10 years as per study procedure.

# 8. End of Trial Definition

This teaching project will be held on one day, participants will be followed up at 6 months following the training to repeat the post-training assessment. This will signal the end of the study.

# 9. Statistical Considerations

# 9.1. Statistical Analysis

Performance characteristics of the participants for diagnosing colonic neoplastic vs. non neoplastic lesions (sensitivity, specificity, NPV, PPV and accuracy) will calculated by comparing predicted histology with actual histology for all polyps and for those diagnosed with high confidence. These performance characteristics between the two groups (face to face classroom training vs. self-training module ) will be compared using the Fisher's ex- act test. A P value of <0.05 will be considered to be statistically significant. *Kappa* statistic will


be used to determine inter-observer agreement in polyp video classification during the training session.

### 9.1.1. Planned Randomisation Methodology

A Computer-generated randomisation system will allow us to allocate the participants into two teaching groups.

# 9.1.2. Planned Sub Group Analyses

Subgroup analysis will include didactic training vs. computer based self-learning. We will also compare the performance of predicting histology of NICE versus SIMPLE versus BASIC in all observations as well as only taking high confidence predictions. We will compare the inter-observer agreement between NICE, SIMPLE and BASIC.

### 9.1.3. Planned Final Analyses

Final analysis will take place after the initial training day and after the 6-month follow up assessment.

### 9.1.4. Power Calculations

Assuming a non-inferiority trial with one-sided distribution (face-to-face training versus computer based training), and power of 90% the sample size is 375 observations (observation=1 video scored). This falls to 271 observations if 0.80 1-beta error is set. As we will use 60 videos per participants, we would need a minimum of 7 participants in each centre. To minimise any potential errors we aim to recruit 14 participants from each centre (7 randomised to face-to-face training and 7 to the computer group).

# 10. Trial Organisational Structure

There is no trial steering committee needed for this teaching project, The members involved are outlined in the administrative information at the start of this protocol.

#### 10.1. Sponsor

University of Birmingham will be the sponsor for this teaching project.

21 of 27 Version date: 09/01/2018 Page:

#### 10.2. **Trials Office**

This project will be run and conducted by the Institute of Translational Medicine

# 11. Confidentiality and Data Protection

Consent for the holding of participant data and publication of findings will be gained from participants online prior to starting the pre and post training assessments.

# 12. Insurance and Indemnity

The University of Birmingham has in place Clinical Trials indemnity coverage for this trial which provides cover to the University for harm which comes about through the University's, or its staff's, negligence in relation to the design or management of the trial and may alternatively, and at the University's discretion provide cover for non-negligent harm to participants.

### 13. Access to the final trial dataset

Dr Marietta Iacucci, Dr Samuel Smith and Hollie Caulfied will have access to the full data set throughout this study

# 14. Publication Policy

It is intended that the results of the study will be reported and disseminated at international conferences such as the British Society of Gastroenterology annual meeting, the United European Gastroenterology Week (UEGW) and the Digestive Diseases Week (DDW) and in peer-reviewed scientific journals such as Endoscopy, Gastrointestinal Endoscopy and Gut. Results will also be disseminated to the local primary care groups, the Oxford and Wessex 'Gut Club' and also to patients via the endoscopy staff and patient forum.

# 15. Reference List

22 of 27 Training Module Version number: 1.0 Version date: 09/01/2018 Page:

#### References:

- Lieberman D, Moravec M, Holub J et al. Polyp size and advanced histology in patients undergoing colonoscopy screening: implications for CT colonography. Gastroenterology 2008; 135: 1100 – 110,
- Rex DK, Overhiser AJ, Chen SC, Cummings OW, Ulbright TM. Estimation of impact of American College of Radiology recommendations on CT colonography reporting for resection of high-risk adenoma fi ndings. Am J Gastroenterol 2009; 104: 149–53
- 3. Hewett DG, Kaltenbach T, Sano Y, et al. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology 2012;143:599-607
- 4. Hassan C, Pickhardt PJ, Rex DK. A resect and discard strategy would improve costeffectiveness of colorectal cancer screening. Clin Gastroenterol Hepatol 2010; 8: 865 – 869
- 5. Ignjatovic A, East JE, Suzuki N et al. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol 2009; 10: 1171 1178
- 6. McGill SK, Evangelou E, Ioannidis JP et al. Narrow band imaging to differentiate neoplastic and non-neoplastic colorectal polyps in real time: a meta-analysis of diagnostic operating characteristics. Gut 2013; 62: 1704 1713
- 7. Wu L, Li Y, Li Z et al. Diagnostic accuracy of narrow-band imaging for the differentiation of neoplastic from non-neoplastic colorectal polyps: a meta-analysis. Colorectal Dis 2013; 15: 3 11
- 8. Sakamoto T, Matsuda T, Aoki T et al. Time saving with narrow-band imaging for distinguishing between neoplastic and non-neoplastic small colorectal lesions. J Gastroenterol Hepatol 2012; 27: 351–355
- Chiu HM, Chang CY, Chen CC et al. A prospective comparative study of narrow-band imaging, chromoendoscopy, and conventional colonoscopy in the diagnosis of colorectal neoplasia. Gut 2007; 56: 373 –379
- 10. Machida H, Sano Y, Hamamoto Y et al. Narrow-band imaging in the diagnosis of colorectal mucosal lesions: a pilot study. Endoscopy 2004; 36: 1094–8
- 11. Gono K, Obi T, YamaguchiMet al. Appearance of enhanced tissue features in narrow-band endoscopic imaging. J Biomed Opt 2004; 9: 568–77,
- 12. Van den Broek FJ, Reitsma JB, Curvers WL, et al. Systematic review of narrow-band imaging for the detection and differentiation of neoplastic and nonneoplastic lesions in the colon (with videos). Gastrointest Endosc 2009;69:124-35
- 13. Chang CC, Hsieh CR, Lou HY et al. Comparative study of conventional colonoscopy, magnifying chromoendoscopy, and magnifying narrow-band imaging systems in the differential diagnosis of small colonic polyps between trainee and experienced endoscopist. Int J Colorectal Dis 2009; 24:1413–9
- 14. Su MY, Hsu CM, Ho YP, Chen PC, Lin CJ, Chiu CT. Comparative study of conventional colonoscopy, chromoendoscopy, and narrow-band imaging systems in differential diagnosis of neoplastic and nonneoplastic colonic polyps. Am J Gastroenterol 2006; 101: 2711–6
- 15. Hoffman A. et al. Recognition and characterization of small colonic neoplasia with high-defintion colonoscopy using i-scan is as precise as chromoendoscopy. Dig Liver Dis. 2010 Jan;42(1):45-50
- 16. Lee CK et al. Narrow-Band Imaging versus i-scan for the real-time histological prediction of diminutive colonic polyps: a prospective comparative study by using the simple unified endoscopic classification. Gastrointest Endosc. 2011 Sep;74(3):603-9
- 17. Yoshida N et al. Ability of a novel blue laser imaging system for the diagnosis of colorectal polyps. Dig Endosc 2014; 26: 250-8.


- 18. Shimoda R et al. The adenoma miss rate of blue-laser imaging vs. white-light imaging during colonoscopy: a randomized tandem trial. Endoscopy 2017; 49: 186-190
- lacucci M et al. Endoscopy (in press)
- 20. Bisschops R et al. BASIC (BLI Adenoma Serrated International Classification) classification for colorectal polyp characterisation with blue light imaging. Endoscopy 2017 Oct 24. doi: 10.1055/s-0043-121570
- 21. Rogart JN, Jain D, Siddiqui UD et al. Narrow-band imaging without high magnification to differentiate polyps during real-time colonoscopy: improvement with experience. Gastrointest Endosc 2008; 68: 1136-45
- 22. Ladabaum U, Fioritto A, Mitani A et al. Real-time optical biopsy of colon polyps with narrow band imaging in community practice does not yet meet key thresholds for clinical decisions. Gastroenterology 2013; 144: 81-91
- Neumann H et al. Learning curve of virtual chromoendoscopy for the prediction of hyperplastic and adenomatous colorectal lesions : a prospective 2-centre study. Gastrointest Endosc. 2013 Jul;78(1):115-20
- 24. Higashi R, Uraoka T, Kato J, et al. Diagnostic accuracy of narrow-band imaging and pit pattern analysis significantly improved for less experienced endoscopists after an expanded training program. Gastrointest Endosc 2010;72:127-35
- 25. Ignjatovic A, Thomas-Gibson S, East JE et al. Development and validation of a training module on the use of narrow-band imaging in differentiation of small adenomas from hyperplastic colorectal polyps. Gastrointest. Endosc. 2011; 73: 128–33
- Khan T, Cinnor B, Gupta N et al. Didactic training vs. computer-based self-learning in the prediction of diminutive colon polyp histology by trainees: a randomised controlled study. Endoscopy 2017; 14: doi: 10.1055/s-0043-116015

24 of 27 Training Module Version number: 1.0 Version date: Page: 09/01/2018

# Appendices

# Appendix 1.

# NICE classification:

Type 1: Hyperplastic

Colour: same or lighter than background

Vessels: none, or isolated lacy vessels coursing across the lesion

Surface pattern: dark or white spots of uniform size, or homogenous absence of pattern.

Type 2: Adenoma

Colour: browner relative to background (verify colour comes from vessels)

Vessels: brown vessels surrounding white structures

Surface pattern: oval, tubular or branched white structures surrounded by brown vessels.

Type 3: deep submucosal invasive cancer

Colour: brown to dark brown relative to background; sometimes patchy white areas

Vessels: Has area (s) of disrupted or missing vessels

Surface pattern: Amorphous or absent surface pattern

The SIMPLE (Simplified Identification Method for Polyp Labelling during the Endoscopy) classification (lacucci M et al Endoscopy in press) was recently developed with the addition of criteria for Sessile Serrated Adenoma (SSA):

Type 1: Hyperplastic

Surface pattern: Round pit

Vessels: None, isolated lacy

Lesion border: Regular

Type 2a: Sessile serrated adenoma/lesion

Surface pattern: Open/dilated (dark) pit

Vessels: None, isolated lacy

Lesion border: Irregular/indistinctive

25 of 27 Version date: 09/01/2018 Page:

Type 2b: Adenoma

Surface pattern: Not round structure: oval, tubular, branched

Vessels: Thick vessels

Lesion border: Regular

Training Module Version number:1.0 Version date: 09/01/2018 

Training Module Version number:1.0 Version date: 09/01/2018 